CLINICAL TRIAL: NCT07325526
Title: A Phase IIa Double-blind, Placebo-controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 3802876 in Participants With Compensated Cirrhosis Due to Metabolic Dysfunction-Associated Steatohepatitis (MASH)
Brief Title: A Study to Test Whether BI 3802876 is Tolerated in People With Compensated Liver Cirrhosis Due to Metabolic Dysfunction- Associated Steatohepatitis (MASH)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1517-0002; 1111-1313-8064 (Registry Identifier: WHO Registry Identifier)
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- Dose group 1 (Experimental)
  Interventions: Drug: BI 3802876
- Dose group 2 (Experimental)
  Interventions: Drug: BI 3802876
- Dose group 3 (Experimental)
  Interventions: Drug: BI 3802876

INTERVENTIONS:
Drug: BI 3802876 — BI 3802876
  Arms: Dose group 1; Dose group 2; Dose group 3
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This study is open to adults with a type of confirmed liver condition called compensated cirrhosis due to Metabolic Dysfunction-Associated Steatohepatitis (MASH). The purpose of this study is to find out how well a study medicine called BI 3802876 is tolerated in people with this condition. The study looks at how different doses of BI 3802876 are handled by the body. BI 3802876 is being developed to improve liver health in people living with this liver condition.

Participants are put in 3 different dose groups randomly, which means by chance. Participants within a group get BI 3802876 or placebo. Placebo looks like BI 3802876 but does not contain any medicine. Participants have more than twice the chance of receiving BI 3802876 than placebo. The study medicine is given as an infusion into a vein.

Participants are in the study for about half a year. During this time, they visit the study site 12 times. At 2 visits, participants get the study medicine. Doctors collect information on any health problems and take blood samples to check how BI 3802876 is handled by the body. They compare results between the groups.

ELIGIBILITY:
Inclusion Criteria :

* Male or female adults ≥18 to ≤75 years of age at the time of screening, and at least the legal age of consent in countries where it is > 18 years
* Patients meeting criteria for Child-Pugh category A without history of previous decompensation event
* Compensated Metabolic Dysfunction-Associated Steatohepatitis (MASH) cirrhosis diagnosed by 1 of the following:

  * Biopsy (collected during screening or ≤ 5 years* prior to screening) showing cirrhosis (fibrosis stage 4) with steatosis or steatohepatitis.
  * Biopsy (collected during screening or ≤ 5 years* prior to screening) showing cryptogenic cirrhosis.
  * Biopsy showing steatosis or steatohepatitis prior to screening without confirmation of fibrosis stage 4, or current or previous imaging showing steatosis with no liver histology available must meet either one of the following inclusion criteria at screening:

    1. Vibration-controlled transient elastography (VCTE) ≥ 15 kilopascals (kPa) plus 1 of the following, Magnetic Resonance Enterography (MRE) ≥4.2 kPa, platelet count <150,000/μL or imaging techniques (computed tomography (CT) scan and/or Magnetic Resonance Imaging (MRI) and/or Ultrasound) suggestive of cirrhosis.
    2. VCTE measurement ≥ 20 kPa
    3. Enhanced Liver Fibrosis (ELF) score ≥ 10.2 *If biopsy was collected > 365 days prior to screening either criteria a, b or c must be met Further inclusion criteria apply.

Exclusion Criteria :

* Patients with clinically significant portal hypertension defined by any of the following:

  * VCTE ≥25 kPa if the platelets are ≥150,000/μL
  * VCTE ≥20 kPa if platelets are <150,000/μL
  * History of esophageal or gastric varices (Grade ≥1) on endoscopy
  * ELF score ≥11.3
  * Hepatic venous pressure gradient (HVPG) ≥10 mmHg
* Other causes of liver disease based on medical history and/or centralized review of liver histology, including but not limited to alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis [PBC], primary sclerosing cholangitis [PSC], autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1- antitryspin deficiency
* Chronic viral hepatitis parameters that would be considered exclusionary for the participation in this trial are (hepatitis B and C testing will be done at screening visit):

  * Hepatitis B virus (HBV): Past or present hepatitis B infection, including a positive hepatitis B surface antigen (HBsAg) and/or detectable HBV Deoxyribonucleic Acid (DNA).
  * Hepatitis C virus (HCV): patients with positive HCV ribonucleic acid (RNA). Patients treated for hepatitis C must have a negative RNA test at screening and be HCV RNA negative for at least 2 years prior to screening in order to be eligible for the trial.
* History of liver transplantation or patients listed for liver transplantation
* Suspicion, confirmed diagnosis, or history of Hepatocellular Carcinoma (HCC)
* Present or past evidence of decompensating events of liver cirrhosis
* Model for End-Stage Liver Disease (MELD) score > 12, unless due to therapeutic anti-coagulation
* History of significant alcohol consumption (defined as intake of > 210 g/week in males and > 140 g/week in females on average over a consecutive period of more than 3 months) within 1 year prior to screening
* International Normalized Ratio (INR) >1.3 unless due to therapeutic anticoagulants or laboratory error Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2027-03-29 (Estimated); Study Completion 2027-03-29 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any Adverse Events (AEs) | up to 134 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 134 days
Maximum measured concentration of the analyte in serum (Cmax) | up to 134 days
Relative change from baseline in N-terminal type III collagen propeptide (PRO-C3) at week 7 | at baseline, at week 7

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southern California Research Center, Coronado, California
  - Orange County Research Center, Lake Forest, California
  - Pfleger Liver Institute, Los Angeles, California
  - Catalina Research Institute, LLC - Montclair, Montclair, California
  - Velocity Clinical Research, San Diego, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - University of Miami, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Piedmont Healthcare-Atlanta, Atlanta, Georgia
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Centricity Research - Morehead City, Morehead City, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Nashville General Hospital, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Epic Medical Research - Carrollton, Carrollton, Texas
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Epic Medical Research - Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases(in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com